CLINICAL TRIAL: NCT01805843
Title: Pulmonary Vascular Changes in Patients With Chronic Myeloid Leukemia With Second-line Therapy Dasatinib vs. Nilotinib
Brief Title: Pulmonary Vasculopathy Under Second-line Therapy of Chronic Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 24-311 ex 10/11
Record Dates: First submitted 2012-10-10; First posted 2013-03-06 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Pulmonary hypertension; chronic myeloid leukemia; dasatinib; nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Hypertension, Pulmonary | interventions — Caves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA will be retained for later examinations at the Biobank, in case that the patient agrees (extra patient information). The blood samples are taken only during routine tests.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- chronic meloid leukemia: echo, exercise echo, and if indicated, right heart catheter
  Interventions: Other: Echo, exercise echo, and if indicated, right heart catheter

INTERVENTIONS:
Other: Echo, exercise echo, and if indicated, right heart catheter — routine echocardiography and special measurements of the right heart are performed at rest and during exercise

SUMMARY:
Chronic myelogenous leukemia (CML) is a chronic myeloproliferative disorder characterized by a translocation between chromosome 9 and 22, leading to a pathogenic tyrosine kinase signal transduction protein. CML can be treated with tyrosine kinase inhibitors (TKIs), which inhibit BCR/ABL kinase, such as imatinib. In about 20% of CML patients who are treated by imatinib, a complete cytogenetic response cannot be achieved. The other two novel TKIs (dasatinib and nilotinib), achieve higher rates of complete cytogenetic response and they are proposed as second-line therapy for imatinib-resistant patients or for those who do not tolerate imatinib. Dasatinib inhibits BCR/ABL kinase in about >300 times in vitro in more than imatinib and also inhibits several other kinases, including the Src family. Src tyrosine kinase is crucial for potassium channel function in human pulmonary arteries. Imatinib and nilotinib do not inhibit the Src.

Incident cases of precapillary PH have been reported in patients who have CML treated with the dasatinib. Improvements were usually observed after withdrawal of dasatinib.

This study is designed to identify incident cases of dasatinib-associated PH and describe pulmonary vascular changes induced by dasatinib. As comparison population will be patients who receive another second-line TKI (nilotinib).

DETAILED DESCRIPTION:
Doppler echocardiography at rest will be performed in each patient. Patients without exercise capacity limitation an exercise test (Doppler echocardiography with spiroergometry) will be performed. Patients who show elevated SPAP at rest or during exercise (in this study SPAP ≥ 40 mmHg) or with reduced exercise capacity (peak VO2 < 75%) a right heart catheterization (RHC) will be suggested. Additionally for the evaluation of exercise capacity a 6 MWD will be performed. This work- up of patients allows clinical and hemodynamic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic myeloid leukemia under second-line therapy with dasatinib or nilotinib
* written informed consent

Exclusion Criteria:

* Manifest pulmonary hypertension
* significant pulmonary disease
* Left-sided heart failure or diastolic compliance dysfunction +
* Hemodynamic relevant valvular disease
* Systemic arterial hypertension (at rest systolic >150 mmHg, diastolic > 90 mmHg, during exercise > 220 mmHg)
* Severe anemia
* Uncontrolled supraventricular and ventricular arrhythmias
* Myocardial infarction (within the last 12 months)
* Pulmonary embolism (within the last 12 months)
* Recent therapy changes (within the last 12 months)
* Recent major surgeries (within the last 12 months)
* For exercise tests: musculoskeletal diseases which may unable the exercise tests.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with chronic myeloid leukemia under second-line therapy with dasatinib or nilotinib,
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
systolic pulmonary arterial pressure during exercise (50W) | at baseline
  In patients who undergo stressechocardiography: systolic pulmonary arterial pressure (SPAP) at 50W will be measured and the comparison between patients under dasatinib and nilotinib therapy will be performed.

SECONDARY OUTCOMES:
peak VO2 | At baseline
  Mean PAP at rest, mPAP at 50W, peak VO2, 6 minute walk distance (6MWD), N terminal pro brain natriuretic peptide (NT-proBNP) at "dasatinib" vs."nilotinib" patients.
  Changes of SPAP at 50 W, pulmonary vascular resistance (PVR) at rest, changes of mPAP at rest and at 50W, peak VO2, 6 MWD, NT-pro BNP- in patients with dasatinib and nilotinib between the baseline and 6 months after.
change of pulmonary arterial pressure | between baseline and after 6 months
  Changes of SPAP at 50 W, pulmonary vascular resistance (PVR) at rest, changes of mPAP at rest and at 50W, peak VO2, 6 MWD, NT-pro BNP- in patients with dasatinib and nilotinib between the baseline and 6 months after.
Pulmonary vascular resistance | at baseline
  In patients who undergo a RHC: pulmonary vascular resistance (PVR) at rest will be measured and the comparison of patients with dasatinib and nilotinib therapy will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Division of Pulmonology, Graz, Austria